CLINICAL TRIAL: NCT01922206
Title: 2/2-Maternal HIV: Multisite Trial to Assist Disclosure to Children
Brief Title: Maternal HIV: Trial to Assist Disclosure to Children
Acronym: TRACK II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Armistead, Distinguished Professor, Georgia State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: MH094233; 1R01MH094233 (NIH)
Record Dates: First submitted 2013-08-02; First posted 2013-08-14 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: HIV
Keywords: HIV; Maternal Disclosure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait-list Control (No Intervention): Participants in the wait-list control condition will receive a group-based version of the TRACK intervention after their 15-month follow up appointment.
- TRACK Intervention (Experimental): 3-session, individually administered psycho-educational intervention to promote maternal disclosure of HIV status to child
  Interventions: Behavioral: TRACK Intervention

INTERVENTIONS:
Behavioral: TRACK Intervention — TRACK Intervention
  3-session, individually administered psycho-educational intervention to promote maternal disclosure of HIV status to child
  Arms: TRACK Intervention

SUMMARY:
The purpose of this Collaborative R01, under Program Announcement PAR-09-153, is to conduct a full-scale trial of an intervention to assist mothers living with HIV (MLH) with disclosing their serostatus to their young age 6 - 14 year old), well children. A pilot study of the intervention has recently been completed (R01 MH077493) and met its major aims. The basis for development of the pilot intervention was work from three R01s (MH057207, currently Yr. 14) designed to longitudinally assess MLH and their children. Within that work, several studies were conducted on maternal disclosure, suggesting disclosure is difficult, and outcomes for MLH and children could be improved by intervention. The pilot study, known in the community as Teaching, Raising, And Communicating with Kids (TRACK), was based on integrative disclosure theory. Results of the pilot trial indicate that those in the intervention group were six times more likely to disclose their HIV/AIDS status to their child than those in the control group (O.R. 6.33); by the 9-month follow-up 33% of intervention MLH disclosed, compared to only 7.3% of the control group. Perhaps more importantly, the intervention group's emotional functioning and their satisfaction improved significantly following the intervention, compared to the control group. Similarly, child mental health indicators among children of intervention MLH were significantly better than control group children at follow-ups. In this study, TRACK II, we propose to conduct a full-scale trial of the intervention in two sites: (1) Los Angeles county (Site 1, where the pilot trial was conducted), which will include a high proportion of Latina families and a smaller proportion of African-American and White families; and (2) Atlanta, Georgia (Site 2, where the primary consultant on the pilot trial conducts research), which will include a high proportion of Southern African-American families, as well as White families. MLH and their children (N = 440 total; 110 mothers and 110 children per site, n = 220 per site) will be assessed at baseline and at 3, 9, and 15-month follow-ups. MLH will be randomly assigned to the intervention or control. Aims are to:

1. facilitate disclosure of the mothers' HIV status to the children, which will include secondary aims of:

   1. increasing mothers' self-efficacy to disclose and respond to child questions regarding HIV;
   2. reducing mothers' fears regarding disclosure and stigma;
   3. improving maternal knowledge of child development and how to provide appropriate levels of information given the age of the child;
2. improve MLH mental health indicators over time (i.e., depression, anxiety, quality of life);
3. improve child mental health indicators over time (i.e., depression, anxiety, acting out behaviors); and
4. improve family functioning indicators (e.g., cohesion, perceived closeness between mother and child).

ELIGIBILITY:
Inclusion Criteria:

* Mother is HIV+
* ability of mother and child to speak and understand English or Spanish
* child is not HIV+
* Child is 6-14 years old
* Child is unaware of maternal HIV status
* child resides with mother

Exclusion Criteria:

* Mother does not consent
* Child does not assent
* Psychosis of mother or child
* Child diagnosed with depression
* child is developmentally delayed
* Recent or anticipated death in the family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2013-03; Primary Completion 2017-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Disclosure of Maternal HIV status to child | Change in disclosure status between time points 3-, 9-, & 15 month follow ups

SECONDARY OUTCOMES:
Child Mental Health Functioning (Composite measure) | 15- month follow up
  Self and Caregiver reported indicators, including the Child Depression Inventory, Piers-Harris Children's Self-Concept Scale, Penn State Worry Questionnaire

OTHER OUTCOMES:
Maternal Functioning (composite measure) | 15 month follow-up
  CES-D, GAD-7, Health-Related Anxiety Questionnaire, Medical Outcomes Study-Health Self-Report, Alcohol and Drug Assessment
Family functioning (composite measure) | 15 month follow-up
  Cohesiveness, routines, parent-child communication, parent-child relationship quality

CONTACTS AND LOCATIONS:
Overall Officials: Lisa P Armistead, Ph.D., Principal Investigator — Georgia State University; Debra Murphy, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing protocols for the longitudinal data from 220 young children and 220 mothers will be in accordance with NIH Notice of Amendment to A-110, consistent with IRB-approved consent restrictions, and follow Inter-University Consortium for Political and Social Research guidelines for data preparation. Data will be stripped of identifiers and available under signed agreement for: (1) using data only for research; (2) securing date using appropriate technology; and (3) destroying or returning data after analyses. Notice of available data will be on both centers' websites, with data use restrictions.

REFERENCES:
- [Derived] Marelich WD, Ali B, Murphy DA, Schulte MT, Armistead L. Predictors of serostatus nondisclosure in mothers living with human immunodeficiency virus receiving a disclosure intervention: Analysis of a randomized clinical trial intervention arm. Health Psychol. 2024 Sep;43(9):663-672. doi: 10.1037/hea0001390. Epub 2024 Apr 25. PMID 38661649
- [Derived] Schulte MT, Armistead L, Murphy DA, Marelich W. Multisite longitudinal efficacy trial of a disclosure intervention (TRACK) for HIV+ mothers. J Consult Clin Psychol. 2021 Feb;89(2):81-95. doi: 10.1037/ccp0000622. PMID 33705165